CLINICAL TRIAL: NCT05782920
Title: Comparison Between Platelet-rich Plasma (PRP) and Hyaluronic Acid (HA) in the Treatment of Cancer-therapy Related Vulvovaginal Atrophy and Its Impact on Sexual Satisfaction
Brief Title: Management of Cancer Therapy Related Vulvovaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Salma samir, As. Prof, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0201349
Record Dates: First submitted 2023-02-19; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP- treated Group A (Active Comparator): 15 female patients will receive 2 vaginal PRP injections one month apart.
  Interventions: Device: Platelet rich plasma
- PRP-HA treated Group B (Active Comparator): 15 female patients will receive 2 vaginal PRP-non-cross-linked HA injections spaced a month apart.
  Interventions: Device: Platelet rich plasma; Device: non cross-linked hyaluronic acid
- Control Group C (Active Comparator): 15 female patients will receive topical non-cross-linked hyaluronic acid gel applied every three days for 2 months as a control group
  Interventions: Device: topical HA gel

INTERVENTIONS:
Device: Platelet rich plasma — PRP can be considered a concentrate of autologous platelet-derived growth factors with known efficacy in tissue regeneration and wound healing.
  Arms: PRP- treated Group A; PRP-HA treated Group B
Device: non cross-linked hyaluronic acid — HA filling is a known modality for rejuvenation
  Arms: PRP-HA treated Group B
Device: topical HA gel — the standard treatment of vaginal atrophy and dryness
  Arms: Control Group C

SUMMARY:
The goal of this clinical trial is to:

1. evaluate the efficacy of PRP injection and PRP injection mixed with non-cross-linked hyaluronic acid compared to the control group receiving standard therapy with topical non-cross-linked hyaluronic acid gel in the treatment of cancer therapy-induced or worsened vulvovaginal atrophy.
2. To evaluate the impact of vulvovaginal atrophy treatment on the sexual satisfaction of both partners.

Patients will be divided randomly into 3 groups:

Group 1: 15 female patients will receive vaginal PRP injections. Group 2: 15 female patients will receive vaginal PRP injections combined with non-cross-linked hyaluronic acid.

Group 3: 15 female patients will receive topical non-cross-linked hyaluronic acid gel as a control group.

DETAILED DESCRIPTION:
1. The first group will receive two treatment of sub-mucosal PRP injection at the outer 3 cm of the vagina with one month interval in between. (17)
2. The second group will receive two treatment of PRP injection mixed with non-cross linked hyaluronic acid at the outer 3 cm of the vagina with one month interval in between.

9. 3-The third group will receive one applicator (5gm) three times per week of topical hyaluronic acid gel for vaginal application which will be prepared in the faculty of pharmacy for 2 months.

Clinical assessment Patients will be assessed for symptoms and signs of vulvovaginal atrophy (VVA) at baseline, one month, two months, and, three months after the end of treatment.

1. Vulvovaginal atrophy (VVA) symptoms (dryness, dyspareunia) will be assessed on a subjective 10-point scale.

   Also, patient satisfaction with each type of treatment will be assessed with a questionnaire at the end of treatment and they will be asked if they wish to repeat the treatment to maintain effectiveness over time (yes or No).
2. For assessment of VVA signs on physical examination, vaginal health index including assessment of pH, overall elasticity, epithelial mucosa, fluid secretion type, and consistency and moisture will be used as an objective method of evaluation of therapy.
3. Assessment of sexual satisfaction of both male and female partners:

Sexual satisfaction was measured using the Arabic version of the Index of Sexual Satisfaction (ISS) and female sexual function index (FSFI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients have symptoms of VVA (vaginal dryness, burning, itching or dyspareunia)

  * Patients with vaginal health index < 15.
  * All patients have already finished cancer therapy or are on anti-estrogen treatment.
  * Married sexually active
  * Patients who are not receiving any VVA treatment for at least 30 days before starting therapy.

Exclusion Criteria:

* Active or recent history of vulvovaginal inflammation or infection

  * History of vulvar or vaginal cancer.
  * Suspicious lesion in the vulvovaginal area on the gynecological examination

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — females only will be included
Enrollment: 45 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Vulvovaginal atrophy vaginal dryness severity scores | before treatment
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy vaginal dryness severity scores | after 1 month
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy vaginal dryness severity scores | after 2 months
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy vaginal dryness severity scores | 3 months follow up
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy dyspareunia severity scores | before treatment
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy dyspareunia severity scores | after 1 month
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy dyspareunia severity scores | after 2 months
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vulvovaginal atrophy dyspareunia severity scores | 3 months follow up
  scores from 0-10 where 0: no symptoms, 1-3: mild symptoms, 4-6: moderate symptoms, 7-10: severe symptoms
Vaginal health index total score | before treatment
  scores range from 5-25 with lower scores signifying greater atrophy
Vaginal health index total score | after 1 month
  scores range from 5-25 with lower scores signifying greater atrophy
Vaginal health index total score | after 2 months
  scores range from 5-25 with lower scores signifying greater atrophy
Vaginal health index total score | 3 months follow up
  scores range from 5-25 with lower scores signifying greater atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Salma Omar, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hersant B, SidAhmed-Mezi M, Belkacemi Y, Darmon F, Bastuji-Garin S, Werkoff G, Bosc R, Niddam J, Hermeziu O, La Padula S, Meningaud JP. Efficacy of injecting platelet concentrate combined with hyaluronic acid for the treatment of vulvovaginal atrophy in postmenopausal women with history of breast cancer: a phase 2 pilot study. Menopause. 2018 Oct;25(10):1124-1130. doi: 10.1097/GME.0000000000001122. PMID 29738415
- [Derived] Omar SS, Elmulla KF, AboKhadr NA, Badawy AA, Ramadan EN, Hassouna AM, Heikal LA, Arafat WO. Comparable Efficacy of Submucosal Platelet-Rich Plasma and Combined Platelet-Rich Plasma Noncrosslinked Hyaluronic Acid Injections in Vulvovaginal Atrophy: A Cancer Survivorship Issue. J Womens Health (Larchmt). 2023 Sep;32(9):1006-1020. doi: 10.1089/jwh.2023.0144. Epub 2023 Jul 7. PMID 37417970